CLINICAL TRIAL: NCT03376893
Title: The Epidemiology of Silent and Overt Strokes in Adults With Sickle Cell Disease: a Prospective Cohort Study
Brief Title: Epidemiology of Silent and Overt Strokes in Sickle Cell Disease
Acronym: ESCD
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Washington University School of Medicine (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Professor of Pediatrics and Medicine, Vanderbilt University Medical Center
Other Study IDs: 161434
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Anemia, Sickle Cell; Sickle Cell Disease; Stroke; Sickle Cell Thalassemia; Sickle Cell-Beta0-Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SCA with overt stroke: Participants have sickle cell disease and a history of overt stroke.
- SCA with silent stroke: Participants have sickle cell disease and a history of silent stroke.
- SCA with no stroke: Participants have sickle cell disease and no history of stroke.

SUMMARY:
Sickle Cell Disease (SCD) is a rare disease occurring in an estimated 100,000 individuals, often poor and underserved, in the US. Silent and overt strokes contribute significantly to morbidity in adults with SCD, resulting in functional impairment, challenges with school and job performance, and premature death. Five NIH-funded randomized controlled trials have identified therapies to prevent silent and overt strokes in children with SCD, including monthly blood transfusion therapy (for preventing initial and recurrent strokes) and hydroxyurea (for preventing initial strokes). Despite the observation that at least 99% of children with SCD in high-income countries reach adulthood, and approximately 60% of adults will experience one or more strokes (~50% with silent strokes and ~10% with overt strokes), no stroke trials have established therapeutic approaches for adults with SCD. For adults with SCD, inadequate evidence-based guidelines exist for secondary stroke prevention strategies. Applying stroke prevention strategies in children may not be effective for stroke prevention in adults with SCD, particularly given the high rate of co-morbidities. Identifying subgroups of adults with SCD and higher incidence coupled with the contribution of established stroke risk factors in the general population (smoking, diabetes, obesity, renal disease) will provide the requisite data required for the first-ever phase III clinical trials focused on secondary stroke prevention in adults.

DETAILED DESCRIPTION:
In three adult SCD centers, we will conduct a prospective cohort study to test the primary hypothesis that the incidence of infarct recurrence (stroke or silent stroke) or new strokes in adults with silent strokes treated with hydroxyurea will be greater than in those without strokes treated with hydroxyurea. We will test two secondary hypotheses: 1) adults with SCD and silent strokes have cognitive morbidity when compared to adults with SCD without silent strokes, and 2) adults with SCD and strokes receiving regular blood transfusion will have a higher incidence of infarct recurrence than those with SCD without strokes. The aims include Aim 1: Compare the incidence of new overt and silent strokes in adults with SCD and silent strokes to a comparison group of adults without silent strokes or overt strokes. Aim 2: Compare the cognitive morbidity of those with silent strokes and overt strokes to those without strokes. Aim 3: Compare the incidence of new overt and silent stroke in adults with SCD and overt strokes receiving transfusion to adults with SCD without silent or overt strokes treated with hydroxyurea. All clinical information and neuroimaging will be centrally adjudicated with masked and experienced neurology and neuroradiology committees. Data generated after completion of this proposal are critical for developing the first-ever phase III trials for secondary stroke prevention therapies in adults with SCD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with sickle cell disease on hemoglobin analysis and/or other confirmatory documentation of phenotype
2. Patients ≥ 18 years of age
3. Patients followed regularly (at least two visits per year) in the hematology clinics
4. Patients who have demonstrated adherence with follow-up visits for ≥ 3 years
5. Patients willing to be followed prospectively for a minimum of 3.5 years and agree to a standard care exit MRI/MRA of the brain, as well as MRI/MRA every 12 to 18 months or participation in VUMC AHA trial with Dr. Jordan as PI. These are adults with SCA aged 18-40 years at study entry, enrolled with any infarct status (none, SCI or overt stroke) and followed prospectively.
6. Willingness to comply with study protocol, routine clinic visits

Exclusion criteria:

1. Participants judged to be non-compliant by the hematologist based on previous experience in terms of clinic appointments and following advice
2. Participants with contraindications to MRI, including individuals with MRI-incompatible foreign metal objects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patient volunteers from the sickle cell disease clinics of participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adjudication of silent stroke in those with reported history of silent stroke and hydroxyurea therapy | Study enrollment
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether a silent stroke has occurred. Radiologically, silent stroke will be defined as a FLAIR T2W hyperintensity greater than 3 mm, visible in two planes. Neurologically, a silent stroke has no neurological sequelae.
Adjudication of new strokes in those with history of silent stroke and on hydroxyurea therapy | Every 12 to 18 months after enrollment
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether a NEW stroke has occurred since the last exams, and if so, whether it is a silent stroke or overt stroke. Radiologically, silent stroke will be defined as a FLAIR T2W hyperintensity greater than 3 mm, visible in two planes. Neurologically, a silent stroke has no neurological sequelae.
Adjudication of new strokes in those with history of silent stroke and on hydroxyurea therapy | At study exit (at least 3.5 years after enrollment)
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether a NEW stroke has occurred since the last exams, and if so, whether it is a silent stroke or overt stroke. Radiologically, silent stroke will be defined as a FLAIR T2W hyperintensity greater than 3 mm, visible in two planes. Neurologically, a silent stroke has no neurological sequelae.

SECONDARY OUTCOMES:
Cognitive morbidity in those with silent or overt stroke | Study enrollment
  All participants will complete the NIH Toolbox CB. The NIH Toolbox CB allows for the evaluation of several cognitive constructs and yields individual measure scores as well as a composite score. This measure will serve as a baseline for all participants.
Cognitive morbidity in those with silent or overt stroke | Every 12 to 18 months after enrollment
  Participants will complete the NIH Toolbox CB. The NIH Toolbox CB allows for the evaluation of several cognitive constructs and yields individual measure scores as well as a composite score. Results will be compared to the previous measurement(s) to determine if change has occurred.
Cognitive morbidity in those with silent or overt stroke | At study exit (at least 3.5 years after enrollment)
  Participants will complete the NIH Toolbox CB. The NIH Toolbox CB allows for the evaluation of several cognitive constructs and yields individual measure scores as well as a composite score. Results will be compared to the previous measurement(s) to determine if change has occurred.
Adjudication of overt stroke in those with reported history of overt stroke and on transfusion therapy | Study enrollment
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether an overt stroke has occurred.
Adjudication of new strokes in those with history of overt stroke and on transfusion therapy | Every 12 to 18 months after enrollment
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether a NEW stroke has occurred since the last exams, and if so, whether it is a silent stroke or overt stroke. Radiologically, silent stroke will be defined as a FLAIR T2W hyperintensity greater than 3 mm, visible in two planes. Neurologically, a silent stroke has no neurological sequelae.
Adjudication of new strokes in those with history of overt stroke and on transfusion therapy | At study exit (at least 3.5 years after enrollment)
  Based on results of an MRI exam and a neurological exam, performed by a physician, the Neuroradiology Committee and the Neurology Committee will come to consensus on whether a NEW stroke has occurred since the last exams, and if so, whether it is a silent stroke or overt stroke. Radiologically, silent stroke will be defined as a FLAIR T2W hyperintensity greater than 3 mm, visible in two planes. Neurologically, a silent stroke has no neurological sequelae.

CONTACTS AND LOCATIONS:
Overall Officials: Lori C. Jordan, PhD, MD, Principal Investigator — Vanderbilt University Medical Center; Michael R DeBaun, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03376893/Prot_000.pdf